CLINICAL TRIAL: NCT03237715
Title: Unbound Bilirubin Levels in Healthy Term and Late Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Thomas Hegyi, Professor, Rutgers University
Other Study IDs: 1
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast fed cohort
  Interventions: Other: Assessment of unbound bilirubin levels
- Formula fed cohort
  Interventions: Other: Assessment of unbound bilirubin levels

INTERVENTIONS:
Other: Assessment of unbound bilirubin levels — Collection of residual blood for measurement of unbound bilirubin

SUMMARY:
Specific Aim 1: To determine total serum bilirubin (TSB) and unbound bilirubin (Bf) levels in term and late preterm infants during the first week of life.

Specific Aim 2: Measure Bf levels in breast fed and formula fed infants and examine their relationship to unbound fatty acid (FFAu) levels.

Specific Aim 3: To demonstrate that phototherapy results in different changes in TSB and Bf.

ELIGIBILITY:
Inclusion Criteria:

* Term and late-preterm infants admitted to the regular care nursery of Robert Wood Johnson University Hospital will be eligible for the study

Exclusion Criteria:

* Infants suffering from genetic, chromosomal or surgical conditions will be excluded.

Ages: 6 Hours to 7 Days | Sex: All
Age Groups: Child
Study Population: Term and late preterm infants admitted to regular care nursery
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Unbound bilirubin levels in term and late preterm infants | Two years
Unbound bilirubin levels in breast-fed versus formula-fed term and late preterm infants | Two years
Effect of phototherapy on unbound bilirubin levels | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No